CLINICAL TRIAL: NCT00475449
Title: A Randomised Controlled Trial to Compare Coronary Artery Bypass Grafting With Percutaneous Transluminal Coronary Angioplasty and Primary Stent Implantation in Patients With Multi-Vessel Coronary Artery Disease
Brief Title: The Stent or Surgery (SoS) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Medtronic (Industry); Guidant Corporation (Industry); Schneider (Unknown); British Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MREC/98/2/123
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; Stent; coronary artery bypass grafting
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: percutaneous coronary intervention
Procedure: coronary artery bypass grafting

SUMMARY:
This study compared two different methods of restoring blood flow to the heart when there has been a narrowing or blockage in the blood vessels that supply the heart. Currently there are two different ways of restoring blood flow. One is heart surgery where a surgeon operates directly on the heart, through an incision in the breast bone (sternum) and takes segments of the patient's (non-essential) veins or arteries and then uses these to bypass blocked or narrowed segments in the coronary arteries. This way additional blood can be "piped" into the heart muscle wall. The second method is coronary angioplasty with stent implantation. Coronary angioplasty is a non-surgical method performed under a local anaesthetic. During angioplasty a special balloon is advanced to the site of a coronary narrowing, then inflated to make it expand and this action removes the narrowing. This is a more simple and less invasive than surgery but its value has been limited by a tendency for narrowings to reoccur(restenosis) in the six months following the treatment. When this happens a repeat procedure is often performed. To reduce the incidence of restenosis coronary stents are implanted. These are tubular metal scaffold devices that are placed inside a coronary artery at the site of a previous narrowing to help keep the artery open. These devices are usually delivered on an angioplasty balloon and expanded into place.

Both treatments are equally effective at preventing death and subsequent myocardial infarction and most doctors are happy to recommend either option. Angioplasty offers a more simple initial procedure but with a chance of needing a repeat performance. Bypass surgery represents a more significant initial undertaking with a longer recovery and convalescent period but in most cases, provides good relief of symptoms. Patient preference plays an important part in the decision process.

Bypass grafting is currently the therapy most frequently performed world-wide. Angioplasty has a number of important advantages but the need for repeat procedures currently limits its appeal.

Since these trials were performed there have been important advances in angioplasty techniques. Prominent amongst these has been the development and use of Coronary Stents which has been shown (in clinical trials) to reduce the need for repeat procedures after an initial angioplasty. Consequently stent implantation is now in routine use world wide.

If angioplasty is performed with coronary stent implantation then this may reduce the need for repeat procedures and address the principal factor currently limiting the value of this approach. If the results were found to be as good as with bypass grafting then patients could benefit from a shorter hospital stay, a less traumatic operation and a shorter recovery period. We therefore wish to compare the outcomes in patients treated with a) bypass grafting or b) angioplasty with coronary stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patient has typical angina pectoris - stable or unstable symptoms.
* Atherosclerotic coronary artery disease demonstrated with selective coronary angiography with a significant lesion present in at least two of the principal epicardial vessel systems.
* Revascularisation procedure clinically indicated.
* Nominated trial surgeon accepts the patient for CABG.
* Nominated trial interventionist accepts the patient for PTCA and stent.
* At least one identified lesion suitable and targeted for primary stent implantation.
* A procedure for the completion of either revascularisation strategy can be performed within 6 weeks of randomisation.

Exclusion Criteria:

* Previous CABG procedure or other thoracotomy.
* Previous coronary interventional procedure (of any type).
* Intervention on any cardiac valve scheduled for the index revascularisation procedure.
* Excision or other intervention on the myocardium scheduled for the index revascularisation procedure.
* Intervention on the great vessels, carotid arteries or aorta scheduled for the index revascularisation procedure.
* Absent autologous graft material.
* Non-cardiac disease influencing survival.
* Acute myocardial infarction in the 48 hours preceding the proposed revascularisation procedure.
* Participation in any other study that would involve deviation from the routine local management of a revascularisation procedure.
* Allergy to anti-platelet agents in local use.
* Language or other communication barrier.
* Follow-up for two years not possible / Patient unreliable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 988 (Actual)
Dates: Start 1996-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
rates of repeat coronary revascularisation | median 2 years, range 1-4 years

SECONDARY OUTCOMES:
i. Myocardial infarction free survival | median 2 years, range 1-4 years
ii. Death | median 2 and 6 years
iii. Myocardial infarction. (Fatal and non-fatal) | median 2 years, range 1-4 years
iv. Left ventricular function as assessed by 2D echocardiography | median 2 years, range 1-4 years
vi. Functional capacity - subjective by NYHA class | median 2 years, range 1-4 years
vii. Anti-anginal medication requirements | median 2 years, range 1-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Stables, Study Chair — Liverpool Cardiothoracic Centre; Ulrich Sigwart, Study Chair — University Hospital, Geneva; Spencer King, Principal Investigator — Fuqua Heart Centre of Atlanta Piedmont Hospital; John Pepper, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Peter Wahrborg, Principal Investigator — Institute of Stress Medicine; William Weintraub, Principal Investigator — Christiana Centre for Outcomes Research; Jacobus Lubsen, Principal Investigator — Erasmus Medical Centre Rotterdam; Petros Nihoyannopolous, Principal Investigator — Hammersmith Hospitals NHS Trust

REFERENCES:
- [Derived] Booth J, Clayton T, Pepper J, Nugara F, Flather M, Sigwart U, Stables RH; SoS Investigators. Randomized, controlled trial of coronary artery bypass surgery versus percutaneous coronary intervention in patients with multivessel coronary artery disease: six-year follow-up from the Stent or Surgery Trial (SoS). Circulation. 2008 Jul 22;118(4):381-8. doi: 10.1161/CIRCULATIONAHA.107.739144. Epub 2008 Jul 7. PMID 18606919